CLINICAL TRIAL: NCT01525199
Title: Study of Cases and Controls on Diagnosis and Treatment Strategies in Patients With NSCLC With or Without EGFR Mutations.
Brief Title: Diagnosis and Treatment Strategies in Patients With NSCLC With or Without EGFR Mutations.
Acronym: IDENTIFY
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OAR-XXX-2011/1
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Stage IIIB/IV; Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer,; Epidermal Growth Factor Receptor mutation,; Lung cancer,; Lung adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case
- Control

SUMMARY:
The purpose of this trial is to compare the evolution of patients receiving first line treatment for locally advanced or metastatic lung cancer, taking into account if they were requested or not the EGFR mutation test as part of the diagnosis and treatment strategy. There is no assignment to any particular therapeutic strategy.

DETAILED DESCRIPTION:
Study of cases and controls on diagnosis and treatment strategies in patients with NSCLC with or without EGFR mutations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of lung adenocarcinoma, stage IIIb/IV.
* Patients under 1st line treatment against lung adenocarcinoma.

Exclusion Criteria:

* Patients not having the information required by the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from specialized sites; all the participating investigators will be oncologists.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 12 months after the diagnosis of advanced disease
Overall Survival | 12 months after the diagnosis of advanced disease
Number of hospitalizations | 12 months after the diagnosis of advanced disease

CONTACTS AND LOCATIONS:
Locations (17):
- Argentina (17):
  - Research Site, Bahía Blanca, Buenos Aires
  - Research Site, Ciudad de Buenos Aires, Buenos Aires
  - Research Site, Junín, Buenos Aires
  - Research Site, La Plata, Buenos Aires
  - Research Site, Lanús, Buenos Aires
  - Research Site, Lomas de Zamora, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, San Carlos de Bolívar, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Santa Rosa, La Pampa Province
  - Research Site, La Rioja, La Rioja Province
  - Research Site, Mendoza, Mendoza Province
  - Research Site, Gral. Roca, Río Negro Province
  - Research Site, San Luis, San Luis Province
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Santa Fe, Santa Fe Province
  - Research Site, San Miguel de Tucumán, Tucumán Province